CLINICAL TRIAL: NCT02679144
Title: NMTT- Neuroblastoma Maintenance Therapy Trial Using Difluoromethylornithine (DFMO)
Brief Title: Neuroblastoma Maintenance Therapy Trial
Acronym: NMTT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Giselle Sholler (Other)
Collaborators: Beat NB Cancer Foundation (Other); Team Parker for Life (Unknown)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NMTRC014
Record Dates: First submitted 2016-02-04; First posted 2016-02-10 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Eflornithine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Difluoromethylornithine (DFMO) (Experimental): Subjects will receive 730 Days of oral difluoromethylornithine (DFMO) at a dose of 750 mg/m2 ± 250 mg/m2 BID (strata 1, 2, 3, and 4) OR 2500 mg/m2 BID (stratum 1B) on each day of study.
  Interventions: Drug: Difluoromethylornithine (DFMO)

INTERVENTIONS:
Drug: Difluoromethylornithine (DFMO) — Subjects will receive 730 Days of oral difluoromethylornithine (DFMO) at a dose of 750 mg/m2 ± 250 mg/m2 BID (strata 1, 2, 3, and 4) OR 2500 mg/m2 BID (stratum 1B) on each day of study.
  Other Names: eflornithine

SUMMARY:
Difluoromethylornithine (DFMO) will be used in an open label, single agent, multicenter, study for patients with neuroblastoma in remission. In this study subjects will receive 730 Days of oral difluoromethylornithine (DFMO) at a dose of 750 mg/m2 ± 250 mg/m2 BID (strata 1, 2, 3, and 4) OR 2500 mg/m2 BID (stratum 1B) on each day of study. This study will focus on the use of DFMO in high risk neuroblastoma patients that are in remission as a strategy to prevent recurrence.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a pathologically confirmed diagnosis of neuroblastoma, < 30.99 years of age and classified as high risk at the time of diagnosis. Exception: patients who are initially diagnosed as non-high-risk neuroblastoma, but later converted (and/or relapsed) to high risk neuroblastoma are also eligible.
* All patients must be in complete remission (CR):

  1. No evidence of residual disease on scan
  2. No evidence of disease metastatic to bone marrow.
* Specific Criteria by Stratum:

Stratum 1/1B: All patients must have completed standard upfront therapy that replicates treatment which patients who were enrolled on ANBL0032 received, including:

intensive induction chemotherapy and (if feasible) resection of primary tumor, followed by: consolidation with high-dose chemotherapy with stem cell transplant and radiotherapy, followed by: immunotherapy with Ch14.18/IL-2/GM-CSF (dinutuximab) and retinoic acid;.

All subjects on Stratum 1/B must have also met the following criteria:

• A pre-transplant disease status evaluation that met International Neuroblastoma Response Criteria (INRC) for CR (complete response), VGPR (very good partial response), or PR (partial response) for primary site, soft tissue metastases and bone metastases. Patients who meet those criteria must also meet the protocol-specified criteria for bone marrow response prior to transplant as outlined below: No more than 10% tumor involvement (based on total nucleated cellular content) seen on any specimen from a bilateral bone marrow aspirate/biopsy.

Stratum 2: Neuroblastoma that is in first complete remission following standard upfront therapy different from that described for Stratum 1.

Stratum 3: Neuroblastoma that failed to have a response of at least PR following induction chemotherapy and surgical resection of the primary tumor, but that has achieved CR following additional therapy.

Stratum 4: Patients who have achieved a second or subsequent CR following relapse(s).

* Pre-enrollment tumor survey: Prior to enrollment on this study, a determination of mandatory disease staging must be performed:

  * Tumor imaging studies including
  * Bilateral bone marrow aspirates and biopsy
  * This disease assessment is required for eligibility and preferably should be done within 2 weeks prior to enrollment, but must be done within a maximum of 4 weeks before enrollment.
* Timing from prior therapy:

Stratum 1/1B: Enrollment no later than 60 days after completion of upfront therapy, (last dose of cis-retinoic acid) with a maximum of 6 cycles of cis-retinoic acid maintenance therapy.

Stratum 2, 3 and 4: Enrollment no later than 60 days from last dose of the most recent therapy.

* Patients must have a Lansky or Karnofsky Performance Scale score of > 50% and patients must have a life expectancy of ≥ 2 months.
* All clinical and laboratory studies for organ functions to determine eligibility must be performed within 7 days prior to enrollment unless otherwise indicated below.
* Patients must have adequate organ functions at the time of registration:

  * Hematological: Total absolute phagocyte count ≥1000/μL
  * Liver: Subjects must have adequate liver function
  * Renal: Adequate renal function
* Females of childbearing potential must have a negative pregnancy test. Patients of childbearing potential must agree to use an effective birth control method. Female patients who are lactating must agree to stop breast-feeding.
* Written informed consent in accordance with institutional and FDA (food and drug administration) guidelines must be obtained from all subjects (or patients' legal representative).

Exclusion Criteria:

* BSA (Body Surface Area) of <0.25 m2.
* Investigational Drugs: Subjects who are currently receiving another investigational drug are excluded from participation.
* Anti-cancer Agents: Subjects who are currently receiving other anticancer agents are not eligible. Subjects must have fully recovered from hematological and bone marrow suppression effects of prior chemotherapy.
* Infection: Subjects who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
* Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 441 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with event free survival (EFS) during study. | 2 years

SECONDARY OUTCOMES:
Length of time that participants experience Overall Survival (OS) | 7 years
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years
Peak Plasma Concentration (Cmax) | 1 year
  Pharmacokinetic assay
Area under the plasma concentration versus time curve (AUC) | 1 year
  Pharmacokinetic assay
Time to reach Peak Plasma Concentration (Tmax) | 1 year
  Pharmacokinetic assay
Number of participants with ODC (Ornithine decarboxylase) single nucleotide polymorphisms. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer at Atrium Health
Locations (49):
- United States (42):
  - University of Alabama, Children's of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UCSF Benioff Children's Hospital Oakland-, Oakland, California
  - Rady Children's Hospital, San Diego, California
  - Rocky Mountain Pediatric Hematology, Denver, Colorado
  - Connecticut Children's Hospital, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - All Children's Hospital Johns Hopkins Medicine, St. Petersburg, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Augusta University Health, Augusta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - St. Lukes, Boise, Idaho
  - Advocate Aurora Research Institute, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Kentucky Children's Hospital, Lexington, Kentucky
  - Norton Children's Research Institute/Affiliated with University of Louisville School of Medicine, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - University of Massachusetts Medical School Worcester, Worcester, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Langone Health Hassenfeld Children's Hospital, New York, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Randall Children's Hospital, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Monroe Carrell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Dell Children's Blood and Cancer Center, Austin, Texas
  - Children's Medical Center, Dallas, Texas
  - Texas Children's Cancer and Hematology Centers, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (7):
  - Alberta Children's Hospital, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janesway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - UHC Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - CHUQ, Québec, Quebec
  - CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Duke ES, Bradford D, Sinha AK, Mishra-Kalyani PS, Lerro CC, Rivera D, Wearne E, Miller CP, Leighton J, Sabit H, Zhao H, Lane A, Scepura B, Pazdur R, Singh H, Kluetz PG, Donoghue M, Drezner N. US Food and Drug Administration Approval Summary: Eflornithine for High-Risk Neuroblastoma After Prior Multiagent, Multimodality Therapy. J Clin Oncol. 2024 Sep 1;42(25):3047-3057. doi: 10.1200/JCO.24.00546. Epub 2024 Jun 25. PMID 38917371
- See also: Beat Childhood Cancer Consortium Website — http://beatcc.org